CLINICAL TRIAL: NCT07121270
Title: Restorative Early Sleep Treatment After the Emergency Department
Acronym: RESTED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Principal Investigator, Anthony Reffi, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17553-01
Record Dates: First submitted 2025-07-21; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Insomnia; Nightmares Associated With Trauma and Stress; Nightmares; PTSD - Post Traumatic Stress Disorder
Keywords: CBT-I; Nightmares; Insomnia; Trauma; Sleep Education; PTSD; CBT-I&N; Acute Trauma; RCT; Early intervention; Behavioral sleep medicine; Posttraumatic stress; Trauma-induced insomnia; Cognitive behavioral therapy; Prevention
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Combat Disorders; Wounds and Injuries; Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): Cognitive Behavioral Therapy (CBT) is an evidence-based treatment modality that focuses on modifying maladaptive or unhelpful thoughts and behaviors.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia; Behavioral: Cognitive Behavioral Therapy for Insomnia and Nightmares
- Sleep Education (Active Comparator): Sleep Education provides general information on human sleep and sleep hygiene guidelines.
  Interventions: Behavioral: Sleep Education; Behavioral: Sleep Education enhanced with Nightmare Education

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Cognitive Behavioral Therapy for Insomnia (CBT-I) is delivered via 6 weekly 60-min sessions via telemedicine. CBT-I is a multisession treatment approach that focuses on sleep-specific behaviors and thoughts through various methods.
  Arms: Cognitive Behavioral Therapy
Behavioral: Cognitive Behavioral Therapy for Insomnia and Nightmares — Cognitive Behavioral Therapy for Insomnia and Nightmares (CBT-I&N) is a combination of CBT for Insomnia (CBT-I) and Exposure, Relaxation, and Rescripting Therapy used for the treatment of nightmares (ERRT). CBT-I&N is delivered via 6 weekly 60-min sessions via telemedicine and includes the modification of sleep habits, exposure, and progressive muscle relaxation.
  Arms: Cognitive Behavioral Therapy
Behavioral: Sleep Education — Sleep education is delivered via telemedicine via 6 weekly 60-min sessions. These sessions will be focused on psychoeducation on sleep after trauma, including common sleep disturbances that may emerge and sleep hygiene guidelines to minimize these disruptions (e.g., wind-down routine, avoid caffeine).
  Arms: Sleep Education
Behavioral: Sleep Education enhanced with Nightmare Education — Sleep education enhanced with nightmare education will include all the components of normal sleep education, as described above, in addition to normalizing the experience of nightmares after trauma and providing psychoeducation on nightmares. The treatment is provided over 6 weekly 60-min sessions via telemedicine.
  Arms: Sleep Education

SUMMARY:
The goal of this randomized controlled trial is to pilot the virtual delivery of cognitive behavioral therapy for insomnia (CBT-I) and nightmares (CBT-I&N) via telehealth as an early intervention for treating posttraumatic sleep disturbance in acute trauma patients exposed to interpersonal violence.

The main aims are to:

1. Test the acceptability, feasibility, and satisfaction of sleep-focused CBT delivered early after trauma
2. Evaluate the impact of sleep-focused CBT delivered early after trauma on sleep disturbance
3. Evaluate the impact of sleep-focused CBT delivered early after trauma on PTSD symptoms

The investigators will compare CBT-I and CBT-I&N to sleep education control.

Participants will meet with a provider for 6 weekly sessions via telehealth and complete surveys on the participants' symptoms.

DETAILED DESCRIPTION:
Participants will be patients who present to Henry Ford Hospital's Emergency Department within >72hr following a potential trauma.

Eligible patients will be randomized (1:1) to the active treatment condition (CBT-I or CBT-I&N) or to the control condition (sleep education with or without nightmare education).

Patients with insomnia and comorbid nightmares who are randomized to the active treatment condition will be triaged to CBT-I&N, whereas patients with insomnia and comorbid nightmares who are randomized to the control condition will be triaged to receive sleep education + nightmare education. All other patients with insomnia only will be triaged to receive either CBT-I (active) or sleep education (control).

ELIGIBILITY:
Inclusion criteria:

* Michigan residents treated at Henry Ford Hospital
* Fluent in English
* Age 18 years or older
* Presenting to ED following exposure to Criterion A trauma (exposure to actual or threatened death, serious injury, or sexual violence) characterized by interpersonal violence (defined as any victimization experience that involved being intentionally and directly harmed by another individual
* i.e., assault with a weapon, physical assault, or sexual assault
* Qualifying trauma occurred within the past ~72hr
* Hospital Mental Health Risk Screen score ≥ 10 (indicating at-risk for developing mental health problems)
* Patient is not in any other cognitive behavioral treatment with a master's level clinician or above
* Patient is appropriate for outpatient treatment and level of acuity does not require inpatient treatment

Exclusion criteria:

* Presenting to ED for non-interpersonal trauma
* Defined as any experience that does not involve being intentionally and directly harmed by another individual
* i.e., falls, motor vehicle collisions, self-injury or suicide attempt
* Current or past history of schizophrenia or other psychoses based on EMR data
* Current or past PTSD based on EMR data
* Unmanaged mania or bipolar disorder based on EMR data
* Active, untreated substance use disorder based on EMR data other than alcohol use disorder, cannabis use disorder, nicotine use disorder, or tobacco use disorder
* Active suicidality:
* Presented to ED with self-inflicted injury or attempted suicide
* Current suicidal ideation with intent (with or without a specific plan) within past month
* Suicide attempts during the past three months
* Current homicidal ideation
* Active substance withdrawal
* Pregnant
* Evidence of a current or past traumatic brain injury or loss of consciousness due to head injury at the time of trauma based on EMR data
* No cell phone, email address, or stable home address
* Evidence or risk of ongoing traumatic exposure (e.g., domestic violence)
* Adults in police custody or Dept of Correction patients
* Evidence of altered mental status, inability to understand study procedures/risks, or otherwise unable to give informed consent
* Admission to an intensive care unit, admission or surgery, medical instability or hemodynamic compromise
* Currently engaged in cognitive behavioral treatment
* Currently living in a nursing home
* Currently working non-standard shifts (outside the hours 7am - 6pm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Session Attendance | 1-Week Post-Treatment
  Session attendance (# visits attended/# of total visits) ≥ 65% indicates feasibility
Retention Rate | 1-Week Post-Treatment
  Retention rate (# CBT patients who completed ≥ 4 sessions/ # randomized to CBT) ≥ 65% indicates acceptability
Patient Satisfaction | 1-Week Post-Treatment
  Patient satisfaction with the CBT treatments will be assessed using the Client Satisfaction Questionnaire. Each item is rated on a 1-4 scale, with higher scores indicating greater satisfaction. Mean scores ≥ 3 indicate satisfaction.
Change in Insomnia Symptoms (Insomnia Severity Index) | From Pre-Treatment to 1-Week Post-Treatment, 1-Month Post-Treatment, and 3-Months Post-Treatment
  The Insomnia Severity Index (ISI) is a commonly used self-report measure of insomnia symptoms. Scores on the ISI range from 0-28, with a higher score indicating greater insomnia severity.

SECONDARY OUTCOMES:
Change in Nightmare Symptoms (Nightmare Disorder Index) | From Pre-Treatment to 1-Week Post-Treatment, 1-Month Post-Treatment, and 3-Months Post-Treatment
  The Nightmare Disorder Index (NDI) is a commonly used self-report measure of nightmare severity. Scores on the NDI range from 0-20, with a higher score indicating greater nightmare disorder severity.
Change in PTSD Symptoms (PTSD Checklist for DSM-5) | From Pre-Treatment to 1-Week Post-Treatment, 1-Month Post-Treatment, and 3-Months Post-Treatment
  The PTSD Checklist for DSM-5 (PCL-5) is a commonly used self-report measure of PTSD severity. Scores on the PCL-5 range from 0-80, with a higher score indicating greater PTSD severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krakow B, Johnston L, Melendrez D, Hollifield M, Warner TD, Chavez-Kennedy D, Herlan MJ. An open-label trial of evidence-based cognitive behavior therapy for nightmares and insomnia in crime victims with PTSD. Am J Psychiatry. 2001 Dec;158(12):2043-7. doi: 10.1176/appi.ajp.158.12.2043. PMID 11729023
- [Background] Ulmer CS, Edinger JD, Calhoun PS. A multi-component cognitive-behavioral intervention for sleep disturbance in veterans with PTSD: a pilot study. J Clin Sleep Med. 2011 Feb 15;7(1):57-68. PMID 21344046
- [Background] Taylor DJ, Pruiksma KE, Mintz J, Slavish DC, Wardle-Pinkston S, Dietch JR, Dondanville KA, Young-McCaughan S, Nicholson KL, Litz BT, Keane TM, Peterson AL, Resick PA; Consortium to Alleviate PTSD. Treatment of comorbid sleep disorders and posttraumatic stress disorder in U.S. active duty military personnel: A pilot randomized clinical trial. J Trauma Stress. 2023 Aug;36(4):712-726. doi: 10.1002/jts.22939. Epub 2023 Jun 15. PMID 37322836